CLINICAL TRIAL: NCT05038527
Title: ABM/P-15 Bone Graft vs Traditional Bone Graft in Adult Spinal Deformity Surgery - a Randomized Controlled Clinical Trial
Brief Title: ABM/P-15 Bone Graft vs Traditional Bone Graft in Adult Spinal Deformity Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: CeraPedics, Inc (Industry)
Responsible Party: Principal Investigator, Martin Heegaard, PhD student and Medical Doctor, Department of Orthopedic Surgery, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABM/P-15-RH-2021
Record Dates: First submitted 2021-08-26; First posted 2021-09-09 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Spine Deformity; Bone Graft; Complications; Adverse Events
Keywords: Adult Spinal Deformity; Bone graft; ABM/P-15; Spine Surgery

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ABM/P-15 bone graft (Experimental): Group A: Bone graft of anorganic bovine bone mineral coated with a bioactive peptide (ABM/P-15)
  Interventions: Device: ABM/P-15 bone graft
- Standard treatment (No Intervention): Group B: Standard bone graft which is a mix of locally harvested bone and a morselized femoral head (allogenic)

INTERVENTIONS:
Device: ABM/P-15 bone graft — RCT (single blinded) where the patients will be randomized into two groups. One group receiving the standard bone graft which is a mix of locally autologous harvested bone and a morselized femoral head (allogenic) and the other group will receive bone graft of anorganic bovine bone mineral coated with a bioactive peptide (ABM/P-15).
  Arms: ABM/P-15 bone graft

SUMMARY:
The purpose of this prospective trial is to investigate ABM/P-15 bone graft versus traditional bone graft in patients undergoing surgery for Adult Spinal Deformity (ASD) in order to provide better clinical results through faster bone healing, no additional surgeries, fewer complications and thereby increase health-related quality of life.

Main hypotheses:

1. The use of ABM/P-15 bone graft is superior to traditional bone graft treatment regarding the incidence of additional surgeries following index surgery for ASD

   Secondary hypotheses:
2. The investigators expect non-inferiority in patient reported outcome measures in the ABM/P-15 bone graft group compared to the control group
3. The investigators expect non-inferiority in the postoperative fusion rates (bone healing) evaluated on CT scans in the ABM/P-15 bone graft group compared to the control group
4. The investigators expect non-inferiority in postoperative incidence of asymptomatic pseudarthrosis in the ABM/P-15 bone graft group compared to the control group
5. The investigators expect non-inferiority in perioperative complications in ABM/P-15 bone graft group compared to the control group
6. The investigators expect the use of ABM/P-15 bone graft to be cost-efficient compared to the traditional treatment in the control group

DETAILED DESCRIPTION:
2. Description and classification of medical device

i-Factor Peptide Enhanced Bone graftTM: "i-FACTOR Bone Graft is a pure, natural form of hydroxyapatite (anorganic bone mineral or ABM) containing P-15™, a synthetic peptide. It is provided in putty form, comprised of ABM/P-15 particles that are suspended in an inert biocompatible hydrogel. Hydroxyapatite is the major mineral component of bone. P-15 is a fifteen amino acid sequence polypeptide, a portion of Type-I collagen that serves as a biomimetic attachment site for bone cells. The hydrogel carrier (glycerin and carboxymethylcellulose, or CMC) forms the matrix that improves overall the handling characteristics and helps contain the i-FACTOR Bone Graft at the surgical site. The bovine-derived ABM particles within the matrix are radiopaque and sized between 250 and 425 microns. i-FACTOR Bone Graft provides a bone graft substitute that is remodeled into new bone during the natural healing process." The i-Factor Peptide Enhanced Bone graftTM is classified as a CE-marked class III medical device.

i-Factor flex FRTM: "i-FACTOR Bone Graft is a pure, natural form of hydroxyapatite (anorganic bone mineral or ABM) containing P-15, a synthetic peptide. i-FACTOR Flex FR is comprised of ABM/P-15 particles that are suspended in an inert biocompatible carrier, and has been lyophylized (freeze-dried) to form flexible strips. Hydroxyapatite is the major mineral component of bone. P-15 is a fifteen amino acid sequence polypeptide, a portion of Type-I collagen that serves as a biomimetic attachment site for bone cells. The carrier (carboxymethylcellulose, glycerin, and purified silk) forms the matrix that helps contain i-FACTOR Flex FR at the surgical site. The bovine-derived ABM particles within the matrix are radiopaque and sized between 250 and 425 microns. i-FACTOR Flex FR provides a bone graft substitute that is remodeled into new bone during the natural healing process." The i-Factor flex FRTM is classified as a CE-marked class III medical device.

Rationale for the project ASD is associated with excessive pain, severe disability and significantly reduces health-related quality of life. Surgical treatment is often considered the only viable option in patients with severe ASD, although surgery is associated with certain risks. In ASD surgery, the risk of revision surgery due to either postoperative mechanical failure of the implants or pseudarthrosis is common. Although several changes to treatment have been implemented in the last decade, revision surgery is still common and necessary in up to 30% of patients following the index procedure. Therefore, increased attention has been directed towards reducing the risk of pseudarthrosis, and ABM/P-15 bone graft may play a considerable role in preventing that. The effects have previously been described in patients undergoing cervical spinal discectomy with promising results. Promising results has also been found in the treatment of periodontal infrabony defects through enhanced regenerative bone capacity. Furthermore, ABM/P-15 bone graft in combination with locally harvested autograft has shown superiority compared to allogenic bone graft in non-instrumented posterolateral fusion. The use of ABM/P-15 bone graft has, however, not been assessed in patients undergoing long instrumented spinal fusion surgery which is the case in ASD surgery. The ABM/P-15 bone graft will be used as its CE-mark intends.

Literature Since the introduction of iliac crest bone graft (ICBG) in 1958 leading to enhanced spinal fusion rates and lowering the rate of pseudarthrosis, bone grafts have been widely accepted as a supplement to instrumented fusion. Autologous bone graft taken from the iliac crest is often considered "gold standard" in spinal surgery due to its biomechanical properties of osteoconductivity, osteoinductivity, and osteogenesis. Osteoconduction is the combination of the three-dimensional structure of the bone graft and the capability of new bone formation on this particular scaffold. Moreover, availability of growth factors stimulating undifferentiated pluripotent cells into bone-forming cells is known as osteoinduction. Lastly, osteogenetic properties in bone synthesis rely on the continuous contribution of vital and established osteoprogenitor cells. Autologous bone graft consist of all three biomechanical properties however; the supply of is limited. Additionally, the use of autologous bone graft has been associated to potential donor-site complications, forcing surgeons to look for other viable options such as allogenic bone grafts or other alternatives such as demineralized bone matrix ceramics, bone morphogenetic protein, autologous growth factors, stem cell products (allogenic bone graft cellular matrix), synthetic peptides and bioactive peptides. Allogenic bone graft is described as the transfer between two genetically dissimilar individuals of the same species and is the second most transplanted tissue only surpassed by blood transfusions. Allogenic bone graft bears the properties of full osteoconduction, variably osteoinduction but completely lacks osteogenic properties due to loss of cellular elements. However, industrialized allogenic bone grafts, as well as other non-autologous bone grafts, does have some important advantages compared to autologous bone graft including decreased operative time, decreased blood loss, no donor-site morbidity and finally, almost unlimited quantities. The allogenic bone grafts (morselized femoral heads) from local bone banks are naturally with some restrictions to quantities, however; allogenic bone grafts compared to autologous bone grafts are more accessible.

The use of bioactive peptides bone grafts (ABM/P-15), such as "i-FACTOR Peptide Enhanced Bone Graft" (Cerapedics, Inc., Westminister, CO), has shown similar effects in PROMs and even superiority in terms of faster formation of bridging bone within 12 months, compared to the "gold standard" autologous bone grafts. ABM/P-15 bone graft is a composite bone substitute consisting of an anorganic bovine-derived hydroxyapatite matrix (ABM) combined with a synthetic 15 amino acid peptide (P-15). The ABM/P-15 bone graft matrix bears the properties of osteconductivity, osteoinductivity and subsequent osteogenesis. The osteconductive ABM acts as a scaffold for the osteoinductive peptide P-15, acting as a binding site for the α2-β1 integrin (Type I collagen) initiating intra- and extracellular signaling pathways for increased production of growth factors, bone morphogenic proteins (BMP) and cytokines. The increased cell proliferation and differentiation ultimately results in osteogenesis.

In a randomized double-blinded clinical trial, significantly increased fusion rates with the use of ABM/P-15 bone graft combined with locally harvested autograft compared to allogenic bone grafts in non-instrumented spondylolisthesis were reported. However; this did not result in overall improved PROMs in the reported 2-year follow-up period. In a systematic review, the total number of ASD surgeries in Medicare USA increased fourfold between 2000 and 2010 and additionally increasing the total costs of spinal deformity surgeries by a 16-fold from $56 million to $958 million 40. One possible explanation could be the increasing elderly population, possibly leading to increased complications and revision surgeries, imposing a major financial and clinical burden on the health care system. Several other studies also suggests the substantial increase in the frequency and expense of ASD surgery. Given the same effectiveness between two surgical index procedures, the natural choice would be to pick the less expensive procedure. However, transparency of costs (direct cost, indirect cost) may economically benefit the health care system through overall reduced patient cost. In a economic evaluation of perioperative adverse events (AE) associated with spinal surgery, an AE rate of 17.4% accounted for 16% of the total in-hospital cost. Optimally, ABM/P-15 bone grafts could reduce complications, revision surgeries and overall costs per patient.

The use of autograft, allogenic bone grafts, Bone Morphogenic Protein (BMP) etc. have been extensively described in ASD patients, however; the use of the ABM/P-15 bone graft has not yet been assessed in this patient population, despite promising effects in other surgical fields. To our knowledge, only five clinical articles have been published regarding the use of ABM/P-15 bone graft in patients with spinal conditions. Of these five clinical studies, one is an annual 2-year follow-up on a previous RCT study, whereas a second study is the use of ABM/P-15 bone graft compared to allogenic bone grafts in non-instrumented lumbar fusion surgery, leaving three studies undertaken in patients undergoing instrumented spinal fusion surgery. One study (level I evidence) reported in the ABM/P-15 bone graft FDA IDE trial study similar fusion rates compared to autograft in single-level anterior cervical discectomy and fusion (ACDF). Another study (level III evidence) reported similar fusion rates compared to autograft in posterior lumbar interbody fusion (PLIF). Lastly, the third study (level IV evidence) reported satisfactory fusion rates for patients who underwent anterior lumbar interbody fusion (ALIF). Conclusively, our study will be the first to examine the use of ABM/P-15 bone graft both in patients undergoing more than one level of instrumented fusion and in ASD patients. The current findings supplemented with the results of this study will be of significant value, since spinal surgery often involves multiple levels of fusion. Furthermore, our study will merely be the second level I next to the FDA IDE trial study performed in 2016.

The use of ABM/P-15 bone graft has, furthermore, been used in the field of odontology regarding periodontal regeneration. Several studies showed significantly enhanced regenerative bone capacity and provided overall better clinical results in the treatment of periodontal infrabony defects.

4. Main Purposes

In a prospective trial, patients undergoing surgery for Adult Spinal Deformity (ASD) will be randomized into two groups. One group receiving the standard bone graft which is a mix of locally autologous harvested bone and a morselized femoral head (allogenic) and the other group will receive bone graft of anorganic bovine bone mineral coated with a bioactive peptide (ABM/P-15). The following parameters across groups will be assessed:

1. The incidence of revision surgery
2. Patient reported outcome measures (PROMs) preoperatively, at 3 months, at 1-year and 2-year follow-up
3. Evaluation of fusion based on CT-scans at 1-year follow-up

e. Perioperative adverse events f. Cost-effectiveness

Main hypotheses

1. The use of ABM/P-15 bone graft is superior to traditional treatment with a mix of locally autologous harvested bone and a morselized femoral head (allogenic) regarding incidence of revision surgery following index surgery for ASD

   Secondary hypotheses
2. The investigators expect non-inferiority in PROMs in the ABM/P-15 bone graft group compared to the control group
3. The investigators expect non-inferiority in the postoperative fusion rates evaluated on CT scans in the ABM/P-15 bone graft group compared to the control group
4. The investigators expect non-inferiority in postoperative incidence of asymptomatic pseudarthrosis in the ABM/P-15 bone graft group compared to the control group
5. The investigators expect non-inferiority in perioperative adverse events in ABM/P-15 bone graft group compared to the control group
6. The investigators expect the use of ABM/P-15 bone graft to be cost-efficient compared to the traditional treatment in the control group

5. Materials and methods Study design Prospective, single-blinded, randomized, controlled clinical trial at a quaternary specialized spine unit covering all deformity surgery in eastern Denmark.

Methods of analysis A prospective, single-blinded, randomized, controlled clinical, single center study where patients scheduled for elective ASD surgery are randomized to receive either bone grafts of ABM/P-15 or the standard locally harvested autograft combined with allogenic bone graft.

Group A: bone graft of anorganic bovine bone mineral coated with a bioactive peptide (ABM/P-15) mixed with locally harvested bone graft. Will be placed directly on the lamina and or in between transverse processes if no lamina. It will be contained by the muscle layer.

Group B: standard bone-grafting which is a mix of locally harvested bone and a morselized femoral head (allogenic) Patient data will be recorded in RedCap, which will generate a random generic identifier number (ID).

All patients will receive the following examinations at the described time:

Questionnaires (30 min): 14 days prior to surgery, 3 months postop, 1 year postop and 2 years postop

X-rays (30 min): 14 days prior to surgery, 7 days postop, 3 months postop, 1 year postop and 2 years postop

CT-scan (30 min): 1 year postop

Incidence of revision surgery will be defined as revision surgery due to any of the following:

* Implant failure (e.g rod breakage, screw breakage, cage displacement/subsidence)
* Pseudarthrosis assessed by CT-scan

Posterolateral fusion will be defined according to the Lenke fusion grading system (Type A-D). Type A and type B will be defined as having fusion, whereas type C and type D will be defined as non-fusion.

Radiographic signs of pseudarthrosis (in accordance to the above) in combinations with patient reported complaints, including pain, will be defined as symptomatic pseudarthrosis, and asymptomatic pseudarthrosis in cases of radiographic pseudarthrosis without patient reported complaints.

The need for accessory anterior support will be assessed for each individual patient, and utilized through ALIF/PLIF. These patients will receive ABM/P-15 bone graft inside the cage.

Radiographic non-fusion of ALIF/PLIF will be defined as one of the following:

* Lack of substantial sclerotic changes in the recipient bone bed
* Lack of visible bridging bone either through the cage or surrounding it as observed on anterior-posterior or lateral radiographs
* Vertebral body translation of <3 mm on lateral radiographs

Bone graft migration at 3-months follow-up will be evaluated on radiographs. Comparison will be made to the immediate postoperative radiographs.

Statistical analysis:

All statistical analyses will be performed by the primary investigator using R (R Development Core Team, 2011, Vienna).

P < 0.05 will be considered significant.

Patient characteristics

1. Continuous data will be compared using Student's t-test (Gaussian distributed data) or Wilcoxon's sum rank test (non-Gaussian data)
2. Categorical variables will be compared using Chi squared or Fisher's exact test

   Randomization procedure Group A: bone graft of anorganic bovine bone mineral coated with a bioactive peptide (ABM/P-15) Group B: standard bone graft which is a mix of locally harvested bone and a morselized femoral head (allogenic) The cohort will be block randomized (10 in each block) according to the above mentioned two groups. Patients will be informed about the possibility of receiving ABM/P-15 bone graft or standard locally harvested autograft combined with allogenic bone graft. The primary investigator will be responsible for the randomization without bias through block randomization of ten patients in each block. The primary investigator will make ten identical envelopes, five with the text "Group A" and five with the text "Group B". The envelopes will be shuffled, and the surgeon will hereafter be presented the ten envelopes and randomly select one. At the next ASD surgery for a new patient, the surgeon will be presented the remaining nine envelopes. When all ten envelopes have been picked for surgery, ten new ones will be made. This randomizes the selection of bone graft bias-free with a fifty-fifty percent chance of ending in either group A or group B.

   The practical completion and investigation of the study Patients evaluated at a multidisciplinary conference and afterwards scheduled for ASD surgery will be identified in the electronic medical records system (Sundhedsplatformen). Patients eligible for inclusion will at first outpatient visit to plan further final surgery (approx. 2 weeks prior to surgery), be informed about the study both in written form and orally. This information will be given by the primary investigator and/or the spine surgeon in a closed separate room after initial surgery planning. All patients have the right to an assessor to all outpatient visits and also during the written and oral information regarding the clinical study. If the patient wishes to bring an assessor to the information meeting regarding the clinical study, a new appointment can be made 3-10 days prior to the surgery date. Therefore, participating in this study will in no way impact the date of the surgery and further treatment. On the day of surgery, a written informed consent will be obtained should the patient decide to participate in this study. No patient will have less than 48 hours to answer, complied with the Helsinki declaration. After the patient agrees to participate in the study the primary investigator will randomize the patient to receive either ABM/P-15 bone graft or the standard of locally harvested autograft combined with allogenic bone graft according to the above mention section "randomization procedure".

   Deviations from standard treatment There will be no deviations from standard treatment since patients will receive either ABM/P-15 bone graft or the similar standard of locally harvested autograft combined with allogenic bone graft.

   All patients will be treated with a posterior spinal instrumentation and fusion (PSF) procedure and anterior support whenever deemed necessary at the surgeon's discretion. Choice of implants, osteotomies, numbers of levels fused will be decided prior to randomization at the multidisciplinary conference where final indication for surgery is confirmed.

   Cost-effectiveness analysis The overall cost per patient undergoing ASD surgery (incl. pre-, peri- and postoperative costs) can be estimated, using: diagnosis codes, procedural codes incl. supplemental codes in conjunction with data extraction from electronic medical records (Sundhedsplatformen). The total cost is calculated using diagnosis-related group (DRG) rates (this include for example: cystitis, pneumonia etc.).

   In the preoperative phase, the investigators will mainly analyze the ABM/P-15 bone graft (i-FACTOR Peptide Enhanced Bone Graft, Cerapedics) purchase price per patient compared to the cost of allogenic morselized femoral head. Furthermore, the investigators will note if extra clinical controls are required.

   In the perioperative phase the investigators will look at surgery time (incision time), time in theater, personnel involved, use of surgery equipment, planning time, waste time etc.

   The postoperative phase will be divided into cost during admission and cost after discharge from the hospital. Here, the investigators will analyze, in particular, the rate of revision surgery and other adverse events during admission. Additionally, length of hospital stay, complications to surgery, readmission to hospital following discharge, including readmission reason, department, time and length of readmission will be analyzed. Moreover, the investigators will look at the total cost of rehabilitative care and use of pain medication following discharge. All reimbursed prescription medicine is recorded in The Danish National Health Service Prescription Database (DNHSPD). These data will be gathered and analyzed as part of the total cost of rehabilitative care. Finally, information regarding reimbursed physiotherapy will also be gathered and analyzed.

   6. Statistical considerations

   Using:

   - Alpha = 5%

   - Statistical power = 80%

   - Estimated revision rate in the non-intervention group: 30%

   - Estimated revision rate in the intervention group: 15%

   Sample size calculation resulted in a sample size of n = 102 in each group.

   In the study the investigators have planned to include and randomize (block-randomization with 10 in each block) a total of 240 patients. This will secure a high statistical power even if some of the participants should drop out during the study.

   7. Patients The participants of the study will be 240 patients that have been scheduled for elective ASD surgery using the usual indications for ASD at the Spine Unit, Department of Orthopedic Surgery, Rigshospitalet. ASD with indication for surgery will be defined as any spinal procedure requiring posterior instrumented fusion at a minimum of 5 levels to the sacrum.

   Patients who have undergone previous lumbar spine surgery for a degenerative condition will be eligible for inclusion.

   8. Risks, side effects and disadvantages The main risks of ASD surgery involve infection, blood-loss, embolism, paresthesia, paralyses or even death. Based on previous studies with ABM/P-15 bone graft, participation in the present study will not expose the patients to any added risks of these complications.

   Side effects and disadvantages that may occur in this clinical trial study (approved in accordance to the regulation rules of medical devices), will be reported to the "Danish Medicines Agency".

   Radiographs:

   Patients will follow the department's routine regarding long standing radiographs pre- and postoperatively after 1 week, 3, 12 and 24 months.

   The standard procedure at our institution is that patients undergoing surgical treatment for ASD are scheduled for a CT-scan 1-year postoperatively. In the present study, the investigators will use this opportunity and analyze the already planned CT-scans in our study.

   In the written consent form patients are asked (yes:no) in regards of recieving information about the clinical study results as well as any consequences the study might have for the individual patient. In case of any secondary findings on the radiographs, patients who replied "no" on the form will not be informed about these findings. Patients who replied "yes" on the form will be informed about any secondary findings on radiographs and proper treatment will hereafter be initiated. The treatment includes referral to the proper department responsible for treating the specific secondary finding.

   10. Information via electronic medical records (Sundhedsplatformen)

   Variables collected:

   ● Name

   ● CPR-number

   ● Address and phone number
   * Birthdate
   * Sex
   * Diagnosis
   * Lifestyle factors such as alcohol consumption, caffeine intake, smoking habits, weight, height and exercise
   * Comorbidities and a ASA score, including medical treatments (including, but not limited to, hypertension, hypercholesterolemia, diabetes mellitus/HbA1C, dialysis dependence, chronic venous insufficiency, end-stage renal disease, liver disorder, congestive heart failure, osteoporosis, ostemalacia, Paget's disease, disseminated cancer diseases, severe psychiatric diseases)

   All above mentioned information gathered via electronic medical records will be used before patient consent and are essential to the clinical study in terms of the recruitment of patients. This information will hereafter be passed on to the primary investigator.

   All below mentioned information gathered via electronic medical records will be used after patient consent. This information is essential to the clinical study in order to proper analyze differences among patients and thereby, conclude on these findings the differences between the ABM/P-15 bone graft versus the traditional bone graft in Adult Spinal Deformity surgery. This information is in particular of relevance in spine surgery when evaluating differences in bone graft treatment. Furthermore, in order to analyze correlations between the two groups, the investigators believe that the below mentioned information are essential in order to make the correlations analysis.

   ● Previous surgical procedures of the spine (date, type and implants)

   ● Surgical parameters, including blood-loss, surgery time, fluid-replacement therapy, levels of surgery, implant types.

   ● Complications to surgery
   * Adverse events during admission
   * Readmission to hospital following discharge, including readmission reason, department, time and length of readmission
   * Mortality
   * Previously filed patient-reported outcome measures
   * Length of hospital stay

   From phone conversations or outpatient clinic visits the following information are collected:
   * Occupation
   * Current use of pain medication
   * Rehabilitative care (expenditures)

   All radiographs will be analyzed which is the standard procedure for all patients undergoing ASD surgery at our institute.

   After written consent from the patient, the primary investigator and Spine unit, Department of Orthopedic Surgery 6011C, Rigshospitalet, will get direct access to the patient's electronic medical records in order to collect the above mentioned variables as a part of this clinical trial study.

   11. Sensitive patient data All sensitive patient data gathered in this project are protected under "General Data Protection Regulation" and "The Data Protection Act". All data will be anonymized.

   No personally identifiable information will be shared with Cerapedics. Only a gathered anonymized data pool with all patients included could potentially be shared and will in no circumstances include sharing of patient data on individual level. In short, no patient will be identifiable.

   14. Recruitment of patients and informed consent The primary investigator/or surgeon will preoperatively inform potential ASD patients about this scientific study regarding the use of ABM/P-15 bone graft versus locally harvested autograft combined with allogenic bone graft at first outpatient visit to plan further final surgery (approx. 2 weeks prior to surgery). All information regarding the scientific study will be given in a closed separate undisturbed room. The patient has the right to an assessor at the conversation. If the patient wishes to bring an assessor to the information meeting regarding the clinical study, a new appointment can be made 3-10 days prior to the surgery date. Therefore, participating in this study will in no way impact the date of the surgery and further treatment. Patients will be thoroughly informed about this clinical trial, handed the "Participation information", "Before participating" and "Participants rights in a scientific researh project" sheets and all questions regarding the study will be answered to the best of spine surgeons abilities. Furthermore, patients will be informed that no participants will have to have to make a final decision at this time and that cancelation of participation in the study will not influence treatment pre-, peri- or postoperatively. No participants will have less than 48 hours to answer, complied with the Helsinki declaration. However, if the patient agrees to participate in this study by signing a written consent, the primary investigator will inform the surgeon on whether to use ABM/P-15 bone graft or the standard locally harvested autograft and allogenic bone graft on the day of surgery as described. It is the primary investigators responsibility and duty to make sure the above mentioned criteria are met.

   Copies of information and informed consent will be given to subjects in this trial.

   15. Publication of results

   All results, including positive, negative or inconclusive results will be published in peer-reviewed scientific journals. Publications will be done as follows:

   1year follow-up study of the interim results 2year follow-up study of the final results

   16. Ethical considerations The investigators do not expect that patients participating in the study will experience any special side effects or complications directly related to the specific use of ABM/P-15 bone graft.

   Patients in both groups will receive the needed amount of bone graft evaluated by the surgeon. The purpose of giving ABM/P-15 bone graft is to provide better clinical results through faster fusion and higher fusion rates, fewer complications, no additional surgeries and improved overall PROMs postoperatively. There has not been performed any fundamental changes in the overall surgery with this new bone graft type. Additionally, a cost-effectiveness analysis of ABM/P-15 bone graft will be performed and might optimize resources in the health care system. This analysis will have no impact on the treatment of patients in this study.

   The study will not be started until approval from the Scientific Ethical Committee of the Capital Region of Denmark and the Danish Data Protection Agency has been obtained, and it will be registered at clinicaltrials.gov. All patients will receive both oral and written information before informed consent to participate is obtained.

   The significant usefulness of the present study is to gather new knowledge concerning further optimization of clinical result postoperatively from ASD surgeries. Knowledge from our study will benefit society in general and optimize utilization of resources, in terms of best treatment for future patients.

   In case of serious adverse preliminary results, data will be analyzed and if this treatment is found to cause significant critical problems compared to other bone grafts (p<0.05), the study will be ended. This preliminary analysis will be performed after the inclusion of 5% of the patients in order to validate the effect of treatment and adverse events. The study is thus designed to minimize unnecessary risk to the patients.

   17. Information regarding compensation The participants are covered by the Danish Patient Compensation Association.

ELIGIBILITY:
Inclusion Criteria:

* Indication for ASD surgery
* Indication for the use of bone graft
* Age ≥ 18 years old at the date of surgery

Exclusion Criteria:

* ASA ≥ 4
* Formally diagnosed with a disease affecting the bone metabolism or wound healing (severe osteoporosis, osteomalacia, Pagets disease, hyperparathyreoidism etc.)
* Disseminated cancer diseases
* Hypersensitivity to any of the i-FACTOR Peptide Enhanced Bone Graft ingredients
* Smoking, extensive alcohol use or abuse of hallucinating drugs
* Severe liver or kidney disorders
* Pregnancy or breastfeeding patients
* Patients estimated not to be able to understand the information sheet or patients, who do not consent to participate in the study.
* Severe psychiatric diseases
* Ongoing infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of revision surgery | 2 years postoperatively
  Incidence of revision surgery will be defined as revision surgery due to any of the following:
  * Implant failure (e.g rod breakage, screw breakage, cage displacement/subsidence)
  * Pseudarthrosis assessed by CT-scan

SECONDARY OUTCOMES:
Patient reported outcome measures (PROMs) - VAS | Preoperatively, immediate postoperatively, 1 year postoperatively, 2 years postoperatively
  Questionnaire: Visuel analog scale (VAS). Scale 1-10. 1 is no pain, 10 is max pain Minimal clinically important difference (MCID) will be used to assess any difference between groups based on previous reports
Patient reported outcome measures (PROMs) - EQ-5D-3L | Preoperatively, immediate postoperatively, 1 year postoperatively, 2 years postoperatively
  Questionnaire: European Quality of Life Five Dimension with 3 levels (EQ-5D-3L). Each question is scored from 1-3, where 3 is given if there are no problems.
  Values will often be presented as a percentage of the total possible amount. The last question is a scale ranging from 1-100. 1 is worst quality of life, 100 is best quality of life Minimal clinically important difference (MCID) will be used to assess any difference between groups based on previous reports
Patient reported outcome measures (PROMs) - Danespine Deformity Basis | Preoperatively, immediate postoperatively, 1 year postoperatively, 2 years postoperatively
  Questionnaire: Danespine deformity basis. Height and weight, walking ability rangin from normal to bound to the bed. Lastly, the questions is asked why they are undergoing surgery with 5 different options.
  Minimal clinically important difference (MCID) will be used to assess any difference between groups based on previous reports
Patient reported outcome measures (PROMs) - SRS-22 | Preoperatively, immediate postoperatively, 1 year postoperatively, 2 years postoperatively
  Questionnaire: Scoliosis Research Sociely Health-Related Quality of Life Questionnaire with 22 questions (SRS-22).
  Each question is scored from 1-5, where 5 is given if there are no problems. Values will often be presented as a percentage of the total possible amount. Minimal clinically important difference (MCID) will be used to assess any difference between groups based on previous reports
Bone-to-bone fusion assessed on CT scans | 1 year postoperatively
  Posterolateral fusion will be defined according to the Lenke fusion grading system (Type A-D). Type A and type B will be defined as having fusion, whereas type C and type D will be defined as non-fusion [48].
Incidence of asymptomatic pseudarthrosis using CT-scans | 1 year postoperatively
  Radiographic signs of pseudarthrosis (in accordance to the above) in combinations with patient reported complaints, including pain, will be defined as symptomatic pseudarthrosis, and asymptomatic pseudarthrosis in cases of radiographic pseudarthrosis without patient reported complaints.
Perioperative adverse events | Intraoperatively, immediate postoperatively during admission, 1 year postoperatively, 2 years postoperatively
  All adverse events will be noted.
Cost-effectiveness analysis | 2 years postoperatively
  The overall cost per patient undergoing ASD surgery (incl. pre-, peri- and postoperative costs) can be estimated, using: diagnosis codes, procedural codes incl. supplemental codes in conjunction with data extraction from electronic medical records (Sundhedsplatformen). The total cost is calculated using diagnosis-related group (DRG) rates (this include for example: cystitis, pneumonia etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heegaard, MD, Ph.D fellow, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Department of Orthopedics, Spine Unit, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The regulation from data protection regulation and data protection act will always be followed and a permission from data protection agency have been obtained (P-2021-518)

REFERENCES:
- [Background] Glassman SD, Bridwell K, Dimar JR, Horton W, Berven S, Schwab F. The impact of positive sagittal balance in adult spinal deformity. Spine (Phila Pa 1976). 2005 Sep 15;30(18):2024-9. doi: 10.1097/01.brs.0000179086.30449.96. PMID 16166889
- [Background] Good CR, Auerbach JD, O'Leary PT, Schuler TC. Adult spine deformity. Curr Rev Musculoskelet Med. 2011 Dec;4(4):159-67. doi: 10.1007/s12178-011-9101-z. PMID 22021017
- [Background] Bari TJ, Hansen LV, Gehrchen M. Surgical correction of Adult Spinal Deformity in accordance to the Roussouly classification: effect on postoperative mechanical complications. Spine Deform. 2020 Oct;8(5):1027-1037. doi: 10.1007/s43390-020-00112-6. Epub 2020 Apr 11. PMID 32279244
- [Background] Pellise F, Vila-Casademunt A, Ferrer M, Domingo-Sabat M, Bago J, Perez-Grueso FJ, Alanay A, Mannion AF, Acaroglu E; European Spine Study Group, ESSG. Impact on health related quality of life of adult spinal deformity (ASD) compared with other chronic conditions. Eur Spine J. 2015 Jan;24(1):3-11. doi: 10.1007/s00586-014-3542-1. Epub 2014 Sep 14. PMID 25218732
- [Background] Lau D, Clark AJ, Scheer JK, Daubs MD, Coe JD, Paonessa KJ, LaGrone MO, Kasten MD, Amaral RA, Trobisch PD, Lee JH, Fabris-Monterumici D, Anand N, Cree AK, Hart RA, Hey LA, Ames CP; SRS Adult Spinal Deformity Committee. Proximal junctional kyphosis and failure after spinal deformity surgery: a systematic review of the literature as a background to classification development. Spine (Phila Pa 1976). 2014 Dec 1;39(25):2093-102. doi: 10.1097/BRS.0000000000000627. PMID 25271516
- [Background] Smith JS, Klineberg E, Lafage V, Shaffrey CI, Schwab F, Lafage R, Hostin R, Mundis GM Jr, Errico TJ, Kim HJ, Protopsaltis TS, Hamilton DK, Scheer JK, Soroceanu A, Kelly MP, Line B, Gupta M, Deviren V, Hart R, Burton DC, Bess S, Ames CP; International Spine Study Group. Prospective multicenter assessment of perioperative and minimum 2-year postoperative complication rates associated with adult spinal deformity surgery. J Neurosurg Spine. 2016 Jul;25(1):1-14. doi: 10.3171/2015.11.SPINE151036. Epub 2016 Feb 26. PMID 26918574
- [Background] Diebo BG, Shah NV, Boachie-Adjei O, Zhu F, Rothenfluh DA, Paulino CB, Schwab FJ, Lafage V. Adult spinal deformity. Lancet. 2019 Jul 13;394(10193):160-172. doi: 10.1016/S0140-6736(19)31125-0. Epub 2019 Jul 11. PMID 31305254
- [Background] Karstensen S, Bari T, Gehrchen M, Street J, Dahl B. Morbidity and mortality of complex spine surgery: a prospective cohort study in 679 patients validating the Spine AdVerse Event Severity (SAVES) system in a European population. Spine J. 2016 Feb;16(2):146-53. doi: 10.1016/j.spinee.2015.09.051. Epub 2015 Oct 8. PMID 26456809
- [Background] Daubs MD, Lenke LG, Cheh G, Stobbs G, Bridwell KH. Adult spinal deformity surgery: complications and outcomes in patients over age 60. Spine (Phila Pa 1976). 2007 Sep 15;32(20):2238-44. doi: 10.1097/BRS.0b013e31814cf24a. PMID 17873817
- [Background] Pitter FT, Lindberg-Larsen M, Pedersen AB, Dahl B, Gehrchen M. Revision Risk After Primary Adult Spinal Deformity Surgery: A Nationwide Study With Two-Year Follow-up. Spine Deform. 2019 Jul;7(4):619-626.e2. doi: 10.1016/j.jspd.2018.10.006. PMID 31202380
- [Background] Arnold PM, Sasso RC, Janssen ME, Fehlings MG, Smucker JD, Vaccaro AR, Heary RF, Patel AI, Goulet B, Kalfas IH, Kopjar B. Efficacy of i-Factor Bone Graft versus Autograft in Anterior Cervical Discectomy and Fusion: Results of the Prospective, Randomized, Single-blinded Food and Drug Administration Investigational Device Exemption Study. Spine (Phila Pa 1976). 2016 Jul 1;41(13):1075-1083. doi: 10.1097/BRS.0000000000001466. PMID 26825787
- [Background] Emecen P, Akman AC, Hakki SS, Hakki EE, Demiralp B, Tozum TF, Nohutcu RM. ABM/P-15 modulates proliferation and mRNA synthesis of growth factors of periodontal ligament cells. Acta Odontol Scand. 2009;67(2):65-73. doi: 10.1080/00016350802555525. PMID 19031159
- [Background] Yukna RA, Krauser JT, Callan DP, Evans GH, Cruz R, Martin M. Multi-center clinical comparison of combination anorganic bovine-derived hydroxyapatite matrix (ABM)/cell binding peptide (P-15) and ABM in human periodontal osseous defects. 6-month results. J Periodontol. 2000 Nov;71(11):1671-9. doi: 10.1902/jop.2000.71.11.1671. PMID 11128913
- [Background] Yukna RA, Krauser JT, Callan DP, Evans GH, Cruz R, Martin M. Thirty-six month follow-up of 25 patients treated with combination anorganic bovine-derived hydroxyapatite matrix (ABM)/cell-binding peptide (P-15) bone replacement grafts in human infrabony defects. I. Clinical findings. J Periodontol. 2002 Jan;73(1):123-8. doi: 10.1902/jop.2002.73.1.123. PMID 11846193
- [Background] Shaikh MS, Husain S, Lone MA, Lone MA, Akhlaq H, Zafar MS. Clinical effectiveness of anorganic bovine-derived hydroxyapatite matrix/cell-binding peptide grafts for regeneration of periodontal defects: a systematic review and meta-analysis. Regen Med. 2020 Dec;15(12):2379-2395. doi: 10.2217/rme-2020-0113. Epub 2020 Dec 24. PMID 33356535
- [Background] Queiroz AC, Nobrega PB, Oliveira FS, Novaes AB Jr, Taba M Jr, Palioto DB, Grisi MF, Souza SL. Treatment of intrabony defects with anorganic bone matrix/p-15 or guided tissue regeneration in patients with aggressive periodontitis. Braz Dent J. 2013;24(3):204-12. doi: 10.1590/0103-6440201302169. PMID 23969907
- [Background] Barros RR, Novaes AB Jr, Roriz VM, Oliveira RR, Grisi MF, Souza SL, Taba M Jr, Palioto DB. Anorganic bovine matrix/p-15 "flow" in the treatment of periodontal defects: case series with 12 months of follow-up. J Periodontol. 2006 Jul;77(7):1280-7. doi: 10.1902/jop.2006.050161. PMID 16805694
- [Background] Mishra PRN, Kolte AP, Kolte RA, Pajnigara NG, Shah KK. Comparative evaluation of open flap debridement alone and in combination with anorganic bone matrix/cell-binding peptide in the treatment of human infrabony defects: A randomized clinical trial. J Indian Soc Periodontol. 2019 Jan-Feb;23(1):42-47. doi: 10.4103/jisp.jisp_339_18. PMID 30692742
- [Background] Fatima G, Shivamurthy R, Thakur S, Baseer MA. Evaluation of anorganic bovine-derived hydroxyapatite matrix/cell binding peptide as a bone graft material in the treatment of human periodontal infrabony defects: A clinico-radiographic study. J Indian Soc Periodontol. 2015 Nov-Dec;19(6):651-8. doi: 10.4103/0972-124X.164766. PMID 26941516
- [Background] Jacobsen MK, Andresen AK, Jespersen AB, Stottrup C, Carreon LY, Overgaard S, Andersen MO. Randomized double blind clinical trial of ABM/P-15 versus allograft in noninstrumented lumbar fusion surgery. Spine J. 2020 May;20(5):677-684. doi: 10.1016/j.spinee.2020.01.009. Epub 2020 Jan 28. PMID 32001384
- [Background] MOE JH. A critical analysis of methods of fusion for scoliosis; an evaluation in two hundred and sixty-six patients. J Bone Joint Surg Am. 1958 Jun;40-A(3):529-54 passim. No abstract available. PMID 13539082
- [Background] Kirzner N, Hilliard L, Martin C, Quan G, Liew S, Humadi A. Bone graft in posterior spine fusion for adolescent idiopathic scoliosis: a meta-analysis. ANZ J Surg. 2018 Dec;88(12):1247-1252. doi: 10.1111/ans.14551. Epub 2018 May 15. PMID 29763982
- [Background] Blanco JS, Sears CJ. Allograft bone use during instrumentation and fusion in the treatment of adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 1997 Jun 15;22(12):1338-42. doi: 10.1097/00007632-199706150-00011. PMID 9201837
- [Background] Kannan A, Dodwad SN, Hsu WK. Biologics in spine arthrodesis. J Spinal Disord Tech. 2015 Jun;28(5):163-70. doi: 10.1097/BSD.0000000000000281. PMID 25978141
- [Background] Giannoudis PV, Dinopoulos H, Tsiridis E. Bone substitutes: an update. Injury. 2005 Nov;36 Suppl 3:S20-7. doi: 10.1016/j.injury.2005.07.029. PMID 16188545
- [Background] Pape HC, Evans A, Kobbe P. Autologous bone graft: properties and techniques. J Orthop Trauma. 2010 Mar;24 Suppl 1:S36-40. doi: 10.1097/BOT.0b013e3181cec4a1. PMID 20182233
- [Background] Kadam A, Millhouse PW, Kepler CK, Radcliff KE, Fehlings MG, Janssen ME, Sasso RC, Benedict JJ, Vaccaro AR. Bone substitutes and expanders in Spine Surgery: A review of their fusion efficacies. Int J Spine Surg. 2016 Sep 22;10:33. doi: 10.14444/3033. eCollection 2016. PMID 27909654
- [Background] Cheng I, Oshtory R, Wildstein MS. The role of osteobiologics in spinal deformity. Neurosurg Clin N Am. 2007 Apr;18(2):393-401. doi: 10.1016/j.nec.2007.01.002. PMID 17556142
- [Background] Mroz TE, Joyce MJ, Lieberman IH, Steinmetz MP, Benzel EC, Wang JC. The use of allograft bone in spine surgery: is it safe? Spine J. 2009 Apr;9(4):303-8. doi: 10.1016/j.spinee.2008.06.452. Epub 2008 Sep 19. PMID 18805063
- [Background] Ehrler DM, Vaccaro AR. The use of allograft bone in lumbar spine surgery. Clin Orthop Relat Res. 2000 Feb;(371):38-45. doi: 10.1097/00003086-200002000-00005. PMID 10693548
- [Background] Arnold PM, Sasso RC, Janssen ME, Fehlings MG, Heary RF, Vaccaro AR, Kopjar B. i-Factor Bone Graft vs Autograft in Anterior Cervical Discectomy and Fusion: 2-Year Follow-up of the Randomized Single-Blinded Food and Drug Administration Investigational Device Exemption Study. Neurosurgery. 2018 Sep 1;83(3):377-384. doi: 10.1093/neuros/nyx432. PMID 28945914
- [Background] Lauweryns P, Raskin Y. Prospective analysis of a new bone graft in lumbar interbody fusion: results of a 2- year prospective clinical and radiological study. Int J Spine Surg. 2015 Feb 3;9:2. doi: 10.14444/2002. eCollection 2015. PMID 25709887
- [Background] Sherman BP, Lindley EM, Turner AS, Seim HB 3rd, Benedict J, Burger EL, Patel VV. Evaluation of ABM/P-15 versus autogenous bone in an ovine lumbar interbody fusion model. Eur Spine J. 2010 Dec;19(12):2156-63. doi: 10.1007/s00586-010-1546-z. Epub 2010 Aug 9. PMID 20694847
- [Background] Axelsen MG, Overgaard S, Jespersen SM, Ding M. Comparison of synthetic bone graft ABM/P-15 and allograft on uninstrumented posterior lumbar spine fusion in sheep. J Orthop Surg Res. 2019 Jan 3;14(1):2. doi: 10.1186/s13018-018-1042-4. PMID 30606209
- [Background] Gomar F, Orozco R, Villar JL, Arrizabalaga F. P-15 small peptide bone graft substitute in the treatment of non-unions and delayed union. A pilot clinical trial. Int Orthop. 2007 Feb;31(1):93-9. doi: 10.1007/s00264-006-0087-x. Epub 2006 Jun 8. PMID 16761146
- [Background] Qian JJ, Bhatnagar RS. Enhanced cell attachment to anorganic bone mineral in the presence of a synthetic peptide related to collagen. J Biomed Mater Res. 1996 Aug;31(4):545-54. doi: 10.1002/(SICI)1097-4636(199608)31:43.0.CO;2-F. PMID 8836852
- [Background] Kubler A, Neugebauer J, Oh JH, Scheer M, Zoller JE. Growth and proliferation of human osteoblasts on different bone graft substitutes: an in vitro study. Implant Dent. 2004 Jun;13(2):171-9. doi: 10.1097/01.id.0000127522.14067.11. PMID 15179094
- [Background] Loenen ACY, Connor J, Johnson S, Davis K, Hannigan N, Barnes T, Arts JJ, van Rietbergen B. Peptide Enhanced Bone Graft Substitute Presents Improved Short-Term Increase in Bone Volume and Construct Stiffness Compared to Iliac Crest Autologous Bone in an Ovine Lumbar Interbody Fusion Model. Global Spine J. 2022 Sep;12(7):1330-1337. doi: 10.1177/2192568220979839. Epub 2021 Jan 7. PMID 33406899
- [Background] Yang XB, Bhatnagar RS, Li S, Oreffo RO. Biomimetic collagen scaffolds for human bone cell growth and differentiation. Tissue Eng. 2004 Jul-Aug;10(7-8):1148-59. doi: 10.1089/ten.2004.10.1148. PMID 15363171
- [Background] Yeramaneni S, Robinson C, Hostin R. Impact of spine surgery complications on costs associated with management of adult spinal deformity. Curr Rev Musculoskelet Med. 2016 Sep;9(3):327-32. doi: 10.1007/s12178-016-9352-9. PMID 27278531
- [Background] Smith JS, Shaffrey CI, Glassman SD, Berven SH, Schwab FJ, Hamill CL, Horton WC, Ondra SL, Sansur CA, Bridwell KH; Spinal Deformity Study Group. Risk-benefit assessment of surgery for adult scoliosis: an analysis based on patient age. Spine (Phila Pa 1976). 2011 May 1;36(10):817-24. doi: 10.1097/BRS.0b013e3181e21783. PMID 20683385
- [Background] McCarthy I, Hostin R, O'Brien M, Saigal R, Ames CP. Health economic analysis of adult deformity surgery. Neurosurg Clin N Am. 2013 Apr;24(2):293-304. doi: 10.1016/j.nec.2012.12.005. Epub 2013 Feb 21. PMID 23561565
- [Background] Raman T, Nayar SK, Liu S, Skolasky RL, Kebaish KM. Cost-Effectiveness of Primary and Revision Surgery for Adult Spinal Deformity. Spine (Phila Pa 1976). 2018 Jun 1;43(11):791-797. doi: 10.1097/BRS.0000000000002481. PMID 29099409
- [Background] Arutyunyan GG, Angevine PD, Berven S. Cost-Effectiveness in Adult Spinal Deformity Surgery. Neurosurgery. 2018 Oct 1;83(4):597-601. doi: 10.1093/neuros/nyx575. PMID 29566174
- [Background] Alvin MD, Miller JA, Lubelski D, Rosenbaum BP, Abdullah KG, Whitmore RG, Benzel EC, Mroz TE. Variations in cost calculations in spine surgery cost-effectiveness research. Neurosurg Focus. 2014 Jun;36(6):E1. doi: 10.3171/2014.3.FOCUS1447. PMID 24881633
- [Background] Hellsten EK, Hanbidge MA, Manos AN, Lewis SJ, Massicotte EM, Fehlings MG, Coyte PC, Rampersaud YR. An economic evaluation of perioperative adverse events associated with spinal surgery. Spine J. 2013 Jan;13(1):44-53. doi: 10.1016/j.spinee.2013.01.003. PMID 23384882
- [Background] Mobbs RJ, Maharaj M, Rao PJ. Clinical outcomes and fusion rates following anterior lumbar interbody fusion with bone graft substitute i-FACTOR, an anorganic bone matrix/P-15 composite. J Neurosurg Spine. 2014 Dec;21(6):867-76. doi: 10.3171/2014.9.SPINE131151. Epub 2014 Oct 17. PMID 25325176
- [Background] Scheer JK, Oh T, Smith JS, Shaffrey CI, Daniels AH, Sciubba DM, Hamilton DK, Protopsaltis TS, Passias PG, Hart RA, Burton DC, Bess S, Lafage R, Lafage V, Schwab F, Klineberg EO, Ames CP; International Spine Study Group. Development of a validated computer-based preoperative predictive model for pseudarthrosis with 91% accuracy in 336 adult spinal deformity patients. Neurosurg Focus. 2018 Nov 1;45(5):E11. doi: 10.3171/2018.8.FOCUS18246. PMID 30453452
- [Background] Ni J, Zheng Y, Liu N, Wang X, Fang X, Phukan R, Wood KB. Radiological evaluation of anterior lumbar fusion using PEEK cages with adjacent vertebral autograft in spinal deformity long fusion surgeries. Eur Spine J. 2015 Apr;24(4):791-9. doi: 10.1007/s00586-014-3745-5. Epub 2015 Jan 25. PMID 25618451
- [Background] Strube P, Hoff E, Hartwig T, Perka CF, Gross C, Putzier M. Stand-alone anterior versus anteroposterior lumbar interbody single-level fusion after a mean follow-up of 41 months. J Spinal Disord Tech. 2012 Oct;25(7):362-9. doi: 10.1097/BSD.0b013e3182263d91. PMID 21716142
- [Background] Brantigan JW, Steffee AD, Lewis ML, Quinn LM, Persenaire JM. Lumbar interbody fusion using the Brantigan I/F cage for posterior lumbar interbody fusion and the variable pedicle screw placement system: two-year results from a Food and Drug Administration investigational device exemption clinical trial. Spine (Phila Pa 1976). 2000 Jun 1;25(11):1437-46. doi: 10.1097/00007632-200006010-00017. PMID 10828927
- [Background] Burkus JK, Gornet MF, Schuler TC, Kleeman TJ, Zdeblick TA. Six-year outcomes of anterior lumbar interbody arthrodesis with use of interbody fusion cages and recombinant human bone morphogenetic protein-2. J Bone Joint Surg Am. 2009 May;91(5):1181-9. doi: 10.2106/JBJS.G.01485. PMID 19411467